CLINICAL TRIAL: NCT05545423
Title: Effect of Instrument-Assisted Soft Tissue Mobilization on Proprioception and Disability in Patients With Cervicogenic Headache: A Parallel Group, Randomized Controlled Trial
Brief Title: Effect of Instrument-Assisted Soft Tissue Mobilization on Proprioception and Disability in Patients With Cervicogenic Headache
Acronym: IASTM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nabil Mahmoud Ismail Abdel-Aal, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/002832
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Cervicogenic Headache
Keywords: instrumented assisted soft tissue mobilization; cervicogenic headache; proprioception
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Intervention Model Description: instrument-assisted soft tissue mobilization and traditional therapy
Who Masked: Investigator, Outcomes Assessor
Masking Description: opaque sealed envelop
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- instrumented assisted soft tissue mobilization (Experimental): patients will receive IASTM three times a week for eight weeks
  Interventions: Other: instrumented assisted soft tissue mobilization; Other: traditional therapy
- traditional therapy (Active Comparator): patients will receive traditional therapy three times a week for eight weeks
  Interventions: Other: traditional therapy

INTERVENTIONS:
Other: instrumented assisted soft tissue mobilization — the appropriate Graston technique instrument will be selected to scan, and then treat the affected area for 30 to 60 seconds per treated area. The procedure will be applied to the superficial cervical fascia and invested the layers of deep cervical fascia that surround all the structures in the neck. Strokes will be applied on the sternocleidomastoids and upper fibers of trapezius muscles. The IASTM technique was applied at a 45° angle in a direction parallel to the treated muscle fibers for 20 seconds, following immediately by an additional 20-seconds application at a 45° angle in a perpendicular direction to the muscle fibers, resulting in a total treatment time of approximately 40 seconds.
  Arms: instrumented assisted soft tissue mobilization
Other: traditional therapy — The exercise program will be in the form of stretching exercises for the sternocleidomastoids (SCM), the scalenes, and upper fibers of trapezius; strengthening isometric exercises for the neck flexors, extensors, lateral flexors, and neck rotators; and postural correction and scapular stabilization exercises

SUMMARY:
This study will be conducted to investigate the effect of instrument assisted soft tissue mobilization technique In pain intensity, frequency of headache, medication Uptake, Suboccipital movement in flexion and extension, rounded shoulder, forward head posture and proprioception of cervical spine in cases of cervicogenic headache related to trigger points and myofascial restrictions when combined with conventional physical therapy modalities.

DETAILED DESCRIPTION:
The International Headache Society has classified the cervicogenic headache as a secondary headache type that is hypothesized to originate due to nociception in the cervical area. The main difference between these patients with and without cervicogenic headache is the lateralization of pressure hyperalgesia to the painful side of the head and neck, there is a unilateral pattern of pressure hyperalgesia in the head and neck that typifies the altered sensory processing in patients with cervicogenic headache. Cervicogenic headache pain has been mostly related to joint, disc and ligament disease of the upper cervical spine. However, the upper cervical nerves also receive afferent inputs from the muscle tissues.

Several physical therapy techniques are proposed for this type of headache. Strength and endurance exercises, when accompanied by stretching exercises, were shown to be an effective treatment for cervicogenic headache patients. The lack of solid evidence of positive effects and risks of serious complications for spinal manipulation should be considered in favor of other physical therapy options associated with less risk. Graston Technique is an instrument assisted soft tissue mobilization (IASTM) treatment method using a tool that generates mechanical micro-traumatic damage to the treated area. It thus creates an inflammatory response to accelerate the healing process and restore flexible, normal tissue. This technique seems to have the therapeutic effects of inhibiting the adhesion of tissue, increasing the number of fibroblasts, and promoting collagen synthesis. eighty patients with carcinogenic headache will be allocated randomly to two equal group. one group will receive IASTM and traditional therapy and other will receive traditional only for eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* 35 to 50 years old
* unilaterality of the head pain
* pain triggered by external pressure over the upper cervical joints (C1-C3)
* pain elicited by the neck movements, and/or sustained awkward positions, reduced neck ROM
* headache intensity pain score of at least 20mm on the Visual Analogue Scale,
* headache frequency of at least once a week for at least 3 months
* minimum neck disability index score of 10 points or greater.

Exclusion Criteria:

* migraine
* tension-type headache
* tumor
* osteoporosis
* fracture
* rheumatoid arthritis and metabolic diseases
* prolonged history of steroid use
* resting blood pressure greater than 140/90 mmHg
* cervical spinal stenosis
* diminished sensation
* central nervous system involvement
* previous head or neck surgery
* whiplash injury history within the last 6 weeks
* head or neck pain treatment within the last month from any practitioner and PT approach for head or neck pain within the last 3 months
* open wounds and psychiatric/cognitive disorders
* patients contraindicated to carotid artery massage

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
joint position error | up to eight weeks
  The Cervical Joint Position Error (JPE) Test is a measurement tool used to clinically assess an individual's cervicocephalic proprioception ability. Cervicocephalic proprioception describes one's sense of position of their head and neck in space. The Cervical JPE Test measures the ability of a blindfolded patient to accurately relocate their head position back to a predetermined neutral point after cervical joint movement. The test is most commonly performed with head movement in the transverse and sagittal planes by cervical range of motion device (CROM).

SECONDARY OUTCOMES:
disability | up to eight weeks
  The neck disability index (NDI) will be used for measuring neck disability and it is a self-patient-completed questionnaire that measures patients' functional status. It contains 10 questions regarding pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation. Each question has six answer choices scored from 0 to 5 as 0 indicates no disability and 5 indicates complete disability. All sections are scored then totaled on a scale from 0 to 50, as zero is the best possible score and 50 is the worst one
headache frequency | up to eight weeks
  the number of days the patients feel headache
headache duration | up to eight weeks
  the total hour of headache
medication intake | up to eight weeks
  from the patient diary in the last week, medication intake will be recorded as follow: 1) not at all; 2) once a week; 3) once every couple of days; 4) once or twice a day; or 5) three or more times a day.
pain intensity | up to eight weeks
  Visual Analogue Scale which is a 100-mm horizontal line will be used for measuring pain intensity. The patients will be instructed to represent their pain intensity level by marking anywhere on the line with "no pain" on the left side and "worst pain" on the right side.
forward head posture | up to eight weeks
  cervical range of motion 2 (CROM2 ruler will be used for assess the forward head posture
rounded shoulder assessment | up to eight weeks
  tape measurement will be used to to assess rounded shoulder: Subjects will be requested to stand normally with their hands hanging beside their bodies to test for rounded shoulder posture. Then, sternal notch, coracoid process, posteriolateral angle of the acromion process and the adjacent thoracic spinous process will be palpated and marked. The distance between sternal notch and coracoid process, and the distance between the posterolateral angle of the acromion process and the adjacent thoracic spinous process will measured by using tape.
suboccipital flexion and extension of cervical vertebra | up to eight weeks
  The cervical range of motion device (CROM) will measure suboccipital flexion and extension of cervical vertebrae. Instruct the subject to position the CROM Instrument as if putting on a pair of glasses. Fasten the velcro strap in line with the bows. Instruct the subject to stand facing away from an outside corner of a wall or edge of an open door frame. The subject's sacrum, thoracic spine, and occiput must be in contact with the corner of the wall or door edge. Instruct the subject to flex the suboccipital area as much as possible while maintaining equal pressure on the skull, thorax, and sacrum. Record this measurement. Instruct the subject to extend the suboccipital area as much as possible without allowing the skull, thorax, and sacrum to leave the contact surface.
headache disability | up to eight weeks
  headache-specific disability questionnaire will be used to assess headache disability. the questionnaire has 9 items. the score for each one from 0 to 10. a score of 10-28% is considered to constitute mild disability; 30-48% is moderate; 50-68% is severe; 72% or more is complete.